CLINICAL TRIAL: NCT00668772
Title: 1-yr Study Comparing TioSal Combo Regimens Versus Single Agent Therapies (Spiriva HandiHaler and Salmeterol PE Capsule)
Brief Title: Tiotropium/Salmeterol Inhalation Powder in COPD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.15; 2007-005107-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-04-17; First posted 2008-04-29 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (5):
- Tiotropium/Salmeterol QD (Experimental): Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule
  Interventions: Drug: Tiotropium/Salmeterol
- Tiotropium QD (Active Comparator): Tiotropium Inhalation Powder, hard gelatine capsule (Spiriva®)
  Interventions: Drug: Tiotropium
- Salmeterol BID (Active Comparator): Salmeterol Inhalation Powder, hard PE capsule
  Interventions: Drug: Salmeterol
- Tiotropium/Salmeterol QD + Salmeterol (Active Comparator): Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule, plus Salmeterol Inhalation Powder, hard PE capsule
  Interventions: Drug: Tiotropium/Salmeterol QD + Salmeterol
- Placebo (Placebo Comparator): Placebo Inhalation Powder, hard PE capsule / hard gelatine capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium/Salmeterol — Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule
  Arms: Tiotropium/Salmeterol QD
Drug: Tiotropium/Salmeterol QD + Salmeterol — Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule, plus Salmeterol Inhalation Powder, hard PE capsule
  Arms: Tiotropium/Salmeterol QD + Salmeterol
Drug: Placebo — Placebo Inhalation Powder, hard PE capsule / hard gelatine capsule
  Arms: Placebo
Drug: Salmeterol — Salmeterol Inhalation Powder, hard PE capsule
  Arms: Salmeterol BID
Drug: Tiotropium — Tiotropium Inhalation Powder, hard gelatine capsule (Spiriva®)
  Arms: Tiotropium QD

SUMMARY:
The primary objectives of this study are to assess bronchodilator efficacy as determined by FEV1, the effect on dyspnoea as determined by the BDI/TDI, the effect on health status as determined bt the SGRQ and the effect on COPD exacerbations

ELIGIBILITY:
Inclusion criteria:

Main:

Diagnosis of COPD Post-bronchodilator FEV1<80% predicted and FEV1/FVC<70% predicted

Exclusion criteria:

Main:

Significant other diseases then COPD Recent MI Any unstable or life-threatening cardiac arrythmia requiring intervention or change in drug therapy during the past year Hospitalisation for cardiac failure during the past year History of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2008-11-21 (Actual); Study Completion 2008-11-21 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response | 12 Weeks, 24 Weeks and 48 Weeks
FEV1AUC 0 8hr response | 12 Weeks, 24 Weeks and 48 Weeks
Mahler TDI focal score | 12 Weeks, 24 Weeks and 48 Weeks
SGRQ total score | 12 Weeks, 24 Weeks and 48 Weeks
Time to first moderate to severe COPD exacerbation | 12 Weeks, 24 Weeks and 48 Weeks

SECONDARY OUTCOMES:
Trough FEV1 response | 4, 36 and 48 weeks
FEV1 AUC0-8h response | 4, 36 and 48 weeks
Peak FEV1 response | 12, 24, 36 and 48 weeks
Use of rescue medication (weekly mean number of puffs of as-needed salbutamol/albuterol per day, daytime and night-time) | 24 hours
Weekly mean number of COPD related night time awakenings | 1 week
FVC (forced vital capacity) AUC0-8h and trough FVC response | 48 weeks
Individual FEV1, FVC and PEF measurements | 48 weeks
Weekly mean morning pre-dose and evening pre-dose PEFs (peak expiratory flow) and FEV1 (recorded by AM2+); PEFs determined by spirometry ] | 48 weeks
Mahler TDI focal score | 4, 36 and 48 weeks
Mahler Dyspnoea Indices (Functional Impairment, Magnitude of Task and Magnitude of Effort) | 4, 12, 24, 36 and 48 weeks
SGRQ total score, and the impact, activity and symptoms domain scores from the SGRQ | 4, 12, 36 and 48 weeks
All adverse events | 48 weeks
Vital signs: pulse rate and blood pressure | Baseline and 4 weeks
Routine blood chemistry, haematology and urinalysis | Baseline and 48 weeks
Vital status of randomised patients | 48 weeks
Number of days in hospital (including ambulance transportation | 48 weeks
Number of unscheduled health care provider visits | 48 weeks
Number of visits in emergency room (including ambulance transportation) | 48 weeks
Number of days in intensive care unit | 48 weeks
Concomitant medications (for instance antibiotics and systemic steroids) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (64):
- United States (16):
  - 1184.15.01069 Boehringer Ingelheim Investigational Site, Anniston, Alabama
  - 1184.15.01071 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1184.15.01054 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1184.15.01063 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1184.15.01064 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1184.15.01065 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1184.15.01052 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1184.15.01055 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1184.15.01058 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1184.15.01062 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1184.15.01072 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 1184.15.01053 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1184.15.01070 Boehringer Ingelheim Investigational Site, New York, New York
  - 1184.15.01057 Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - 1184.15.01059 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1184.15.01051 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Austria (2):
  - 1184.15.43052 Boehringer Ingelheim Investigational Site, Gänserndorf
  - 1184.15.43053 Boehringer Ingelheim Investigational Site, Vienna
- Canada (8):
  - 1184.15.02057 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1184.15.02059 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1184.15.02055 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1184.15.02058 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1184.15.02051 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 1184.15.02053 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1184.15.02060 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1184.15.02056 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Denmark (4):
  - 1184.15.45054 Boehringer Ingelheim Investigational Site, Aalborg
  - 1184.15.45052 Boehringer Ingelheim Investigational Site, Kolding
  - 1184.15.45051 Boehringer Ingelheim Investigational Site, Odense C
  - 1184.15.45053 Boehringer Ingelheim Investigational Site, Silkeborg
- Estonia (2):
  - 1184.15.37252 Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - 1184.15.37251 Boehringer Ingelheim Investigational Site, Tallinn
- Finland (2):
  - 1184.15.35852 Boehringer Ingelheim Investigational Site, Oulu
  - 1184.15.35851 Boehringer Ingelheim Investigational Site, Tampere
- France (3):
  - 1184.15.3350A Boehringer Ingelheim Investigational Site, Marseille
  - 1184.15.3351A Boehringer Ingelheim Investigational Site, Nantes
  - 1184.15.3352A Boehringer Ingelheim Investigational Site, Paris
- Germany (5):
  - 1184.15.49056 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1184.15.49053 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1184.15.49057 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1184.15.49052 Boehringer Ingelheim Investigational Site, Hanover
  - 1184.15.49058 Boehringer Ingelheim Investigational Site, Hanover
- Hungary (4):
  - 1184.15.36055 Boehringer Ingelheim Investigational Site, Deszk
  - 1184.15.36053 Boehringer Ingelheim Investigational Site, Érd
  - 1184.15.36054 Boehringer Ingelheim Investigational Site, Szarvas
  - 1184.15.36052 Boehringer Ingelheim Investigational Site, Szeged
- 1184.15.39051 Boehringer Ingelheim Investigational Site, Florence, Italy
- Latvia (3):
  - 1184.15.37154 Boehringer Ingelheim Investigational Site, Balvi
  - 1184.15.37152 Boehringer Ingelheim Investigational Site, Jelgava
  - 1184.15.37153 Boehringer Ingelheim Investigational Site, Tukums
- 1184.15.37053 Boehringer Ingelheim Investigational Site, Klaipėda, Lithuania
- Netherlands (3):
  - 1184.15.31051 Boehringer Ingelheim Investigational Site, Breda
  - 1184.15.31054 Boehringer Ingelheim Investigational Site, Utrecht
  - 1184.15.31052 Boehringer Ingelheim Investigational Site, Zutphen
- Slovakia (2):
  - 1184.15.42153 Boehringer Ingelheim Investigational Site, Bratislava
  - 1184.15.42154 Boehringer Ingelheim Investigational Site, Bratislava
- South Africa (3):
  - 1184.15.27051, Bellville
  - 1184.15.27052, Cape Town
  - 1184.15.27053, Somerset West
- South Korea (3):
  - 1184.15.82051 Boehringer Ingelheim Investigational Site, Jeonju
  - 1184.15.82052 Boehringer Ingelheim Investigational Site, Suwon
  - 1184.15.82053 Boehringer Ingelheim Investigational Site, Wŏnju
- Sweden (2):
  - 1184.15.46053 Boehringer Ingelheim Investigational Site, Boden
  - 1184.15.46051 Boehringer Ingelheim Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/